CLINICAL TRIAL: NCT06331065
Title: Promoting Mental Health at Work Among Hospital Professionals: Implementation and Evaluation of the Effects of an Intervention Based on Mindfulness Meditation in the Workplace - PROMIND Study
Brief Title: Promoting Mental Health at Work Among Hospital Professionals
Acronym: PROMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_1180; ID-RCB (Other: 2023-A01756-39)
Record Dates: First submitted 2024-02-21; First posted 2024-03-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Issue
Keywords: mindfulness; prevention; psychological fulfilment; realistic assessment; occupational health promotion; mental health at work; pilot study; healthcare workers
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness meditation practice group (Experimental): Group informed about mindfulness meditation and experimenting with an adapted program based on mindfulness meditation (intervention group).
  Interventions: Other: Information session on mindfulness meditation and questionnaires; Device: Mindfulness meditation experimentation, practice program, questionnaires, individual interview and focus group
- Group without mindfulness meditation practice (Active Comparator): Group informed about mindfulness meditation and without experimentation of mindfulness meditation practice (control group).
  Interventions: Other: Information session on mindfulness meditation and questionnaires

INTERVENTIONS:
Other: Information session on mindfulness meditation and questionnaires — The information session on mindfulness meditation is an information meeting on the PROMIND study opened to all hospital professionals from the 8 participating departments, i.e. the intervention and control groups.
  During this information session, it is specified that it is desirable for the non-intervention groups to maintain their usual practice (or non-practice) during the study, without starting a new practice of mindfulness meditation.
  Before this meeting, the baseline questionnaires are administered. Immediately after this time, the questionnaire on representations of mindfulness meditation is administered.
Device: Mindfulness meditation experimentation, practice program, questionnaires, individual interview and focus group — After randomization, a mindfulness meditation trial session is offered to all professionals in the intervention group follow by the questionnaire on representations of mindfulness meditation administration.
  Then, interdepartmental focus groups is conducted with leaders. The following mindfulness meditation program consists of 10 1-hour sessions within 15 days, in groups of up to 15 professionals, conducted at the participants' place and time of work, by a certified mindfulness meditation trainer with a recommended daily practice of 10-20 minutes with the possibility of a longer duration, and an audio guidance tool adapted to the study.
  After the program, and 3 months later, questionnaires are administered for both groups.
  For the intervention group, individual interviews, and inter-departmental focus groups (leaders) are carried out at the end of the intervention, and intra-departmental focus groups are conducted 3 months after the end.
  Arms: Mindfulness meditation practice group

SUMMARY:
Mental health is a state of well-being in which a person can realize his/her potential, cope with the normal stresses of life, work productively and contribute to his/her community. It refers to a continuum that extends from the promotion of well-being and the prevention of mental disorders to the treatment and rehabilitation of people suffering from these disorders.

Healthcare professionals face major mental health challenges, due to the demands of their profession, which is characterized by heavy workloads and confrontation with human distress. The frequency of mental health problems among hospital staff is high, at all stages (malaise, distress, pathologies). A meta-analysis found that caregivers suffer from around 30% anxiety, 30% depression, 30% psychotrauma and 45% sleep disorders.

According to the French Labor Code, employers are responsible for the physical and mental health of their employees. The Hospices Civils de Lyon establishment project includes a section on the prevention of psycho-social risks, quality of working life and management.

Healthcare professionals, like the general population, have high expectations of non-medication treatments. These non-medication interventions aim to prevent, treat, or cure a health problem. They are non-invasive and non-pharmacological, with certain observable impacts supported by scientific evidence.

Mindfulness meditation is one of the most extensively studied non-medication interventions in mental health. Declined in different modalities, its effects focus on improving resilience with efficacy on physical and mental well-being (stress, anxiety, burnout, affect), and their physiological corollary (cardiac and respiratory rhythms), acceptance of reality in stressful situations, reduced interpersonal conflict in emergencies and, more broadly, impact on relational behaviours (anti- and pro-social), teamwork. Managers also benefit, with a strengthening of the aspiration to lead, in a vision fully at the disposal of others.

Mindfulness meditation appears to be a practice that promotes mental well-being and could contribute to fulfilment at work.

The challenge is to offer a mindfulness meditation program in a hospital department for individual and collective benefit.

The main objective is to evaluate the evolution of psychological fulfilment in the workplace of hospital healthcare professionals in a 5-month meditation program between the baseline and the end of the program, in comparison with the evolution over the same period of a control group.

The expected outcome is to show that it is possible to implement a mindfulness meditation intervention for hospital staff in care departments, whatever their status or profession, with individual and collective benefits for mental health, psycho-social risks (stress, violence, etc.) and work organization. If it proves to be effective and acceptable, this intervention could be offered more widely within the institution and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Being a Hospices Civils de Lyon professional working in a department participating in the project
* Being of legal age
* Having given written consent including voice recording for focus groups and semi-structured interviews

Exclusion Criteria:

* Self-reported neuro-psychiatric pathology with current severe clinical instability
* Adults under legal protection (guardianship, curators)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Persons unable to understand or write in French
* Pregnant and nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Psychological fulfilment at work | Baseline: before the intervention and immediately after the intervention
  Self-reported psychological fulfilment at work questionnaire for the intervention and control groups.
  13-item questionnaire validated in French. Each item is scored 1-7 (1 = strong disagreement; 7 = strongly agree), yielding a total between 13 and 91 (a high score indicating a high level of psychological fulfillment at work).

SECONDARY OUTCOMES:
Psychological fulfilment at work | 3 months immediately after the end of the intervention
  Self-reported psychological fulfilment at work questionnaire for the intervention and control groups.
  13-item questionnaire validated in French. Each item is scored 1-7 (1 = strong disagreement; 7 = strongly agree), yielding a total between 13 and 91 (a high score indicating a high level of psychological fulfillment at work).
Mindful state | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on the mindful state measured by the Five Facet Mindfulness Questionnaire (15 items) (FFMQ-15).
  Each item is scored on a 5-point Likert scale (1 = never or very rarely true; 2 = rarely true; 3 = sometimes true; 4 = often true; 5 = very often or always true).
  Higher scores mean a more mindful state.
Aggressiveness | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on aggressiveness measured by the 12-item Aggression Questionnaire (AQ12).
  Each item is scored from 1 to 6 (1 = not me at all; 6 = quite me). Higher scores mean a higher level of aggressiveness.
Impulsivity, experience of being disturbed by conflict, and psychological safety. | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on impulsivity, experience of being disturbed by conflict, patient support, and psychological safety measured by a visual analog scale (VAS).
  The VAS ranges from "not at all" (0) to "completely" (10). Higher scores mean a greater impulsivity, a greater experience of being disturbed by conflict and a greater psychological safety.
Occupational stress | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on occupational stress measured by the Job content questionnaire (26 items) Each item is scored from 1 to 4 on a 4-point Likert scale (1 = strongly disagree; 2 = disagree; 3 = agree; 4 = strongly agree).
  The higher the scores, the higher the levels of occupational stress.
Collective activity | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on collective activity ameasured with 4 items by self-assessment using a visual analog scale (VAS).
  Each item is scored from 0 to 10 (0 = strongly disagree; 10 = strongly agree). A higher score indicating greater collective activity.
Organizational leeway | Baseline: before the intervention, immediately after the intervention and 3 months immediately after the intervention
  Intervention's impact on organizational leeway measured by a a visual analog scale (VAS).
  Item 1 is scored with a 5-point VAS (always; most of the time; sometimes; rarely; never). Item 2 is score with a 4-point VAS (never; sometimes; often; always). Items 3 and 4 are scored from 0 to 5 (0 = strongly disagree; 5 = strongly agree).
  A high frequency on item 1, a low frequency on item 2, a low score on item 3 and a high score on item 4 each indicate higher organizational leeway.
Evolution of participants' representation of mindfulness meditation | Before and after the information session on mindfulness meditation, immediately after the first experimental session, immediately after the program and 3 months after the program
  The evolution of participants' representation of mindfulness meditation is measured by Devilly and Borkovec's adapted credibility and expectations questionnaire (6 items).
  Items 1 (I), 2 (I), 3 (I) and 1 (II) are scored from 1 to 9 (1 = not at all consistent /helpful /confident; 9 = very consistent /helpful /confident) and items 4 (I) and 2 (II) are scored from 0% to 100%. An expectancy score is provided by items 4 (I), 1 (II) and 2 (II). A credibility score is provided by items 1 (I), 2 (I), and 3 (I). Higher scores indicate higher levels of expectancy and credibility.
The representation of mindfulness meditation among professionals | Before the program, up to 12 months , 1 and 3 months after the end of the intervention
  Description of the representation of mindfulness meditation measured from verbatim from focus groups.
The representation of mindfulness meditation among professionals | 1 and 3 months after the end of the intervention
  Description of the representation of mindfulness meditation measured from semi-structured interviews.
The representation of mindfulness meditation among professionals | up to 12 months
  Description of the representation of mindfulness meditation measured from verbatim from observation reports.
Fidelity and adherence to the mindfulness meditation intervention | At study completion, an average of 15 months
  Assessing the number of sessions attended, participants and practices in daily life.
Fidelity and adherence to the mindfulness meditation intervention | At study completion, an average of 15 months
  Assessing the duration of the sessions
Barriers and facilitators to the implementation | At study completion, an average of 15 months
  Assessing barriers and facilitators to the implementation through verbatim from focus groups.
Barriers and facilitators to the implementation | At study completion, an average of 15 months
  Assessing barriers and facilitators to the implementation through verbatim from semi-structured interviews.
Mechanisms of the intervention effects | At study completion, an average of 15 months
  Qualitative exploration and description of intervention effects and the mechanisms by which they are produced.
  The objective and methods are open-ended, with no preconceived ideas about the effects produced by the intervention, their mechanisms, and the way in which these mechanisms may be activated (or not) depending on the implementation context. It is based on a triangulation of three complementary methods: 1- non-participant observation.
Mechanisms of the intervention effects | At study completion, an average of 15 months
  Qualitative exploration and description of intervention effects and the mechanisms by which they are produced.
  It is based on a triangulation of three complementary methods: 2- focus groups.
Mechanisms of the intervention effects | At study completion, an average of 15 months
  Qualitative exploration and description of intervention effects and the mechanisms by which they are produced.
  It is based on a triangulation of three complementary methods: 3- semi-structured individual interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Ludivine NOHALES, Study Chair — Hospices Civils de Lyon
Locations (8):
- France (8):
  - Neurology Department, Pierre Wertheimer Hospital (Hospices Civils de Lyon), Bron
  - Pediatric Intensive Care Unit - Continuous Monitoring, Femme Mère Enfant Hospital (Hospices Civils de Lyon), Bron
  - Department of Geriatrics, Edouard Herriot Hospital (Hospices Civils de Lyon), Lyon
  - Neonatology and neonatal intensive care unit, Croix-Rousse Hospital (Hospices Civils de Lyon), Lyon
  - Department of Anesthesia and Intensive Care, Edouard Herriot Hospital (Hospices Civils de Lyon), Lyon
  - Anaesthesia - Intensive Care and Perioperative Medicine Department, Lyon South Hospital (Hospices Civils de Lyon), Pierre-Bénite
  - Department of Physical Medicine and Neurological Rehabilitation, Henry Gabrielle Hospital (Hospices Civils de Lyon), Saint-Genis-Laval
  - Department of Geriatrics, Charpennes Hospital (Hospices Civils de Lyon), Villeurbanne